CLINICAL TRIAL: NCT02789683
Title: Effects of Emulsification and Lipid Droplet Size on Postprandial Metabolic Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2015/00509
Record Dates: First submitted 2016-04-19; First posted 2016-06-03 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Metabolic Diseases
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fine emulsion (Experimental): Emulsion with small lipid droplet size served together with white bread
  Interventions: Other: Fine emulsion
- Coarse emulsion (Experimental): Emulsion with large lipid droplet size served together with white bread
  Interventions: Other: Coarse emulsion
- Control (Experimental): Non-emulsified oil and water served together with white bread
  Interventions: Other: Control

INTERVENTIONS:
Other: Fine emulsion — Emulsion is made up of distilled water, olive oil and emulsifier. Emulsion will be flavored, sweetened (sucralose) and served in a portion of 300ml and approximately 3 slices of white bread (50g of available carbohydrate). Additional glass of plain water will be provided with every treatment.
  Arms: Fine emulsion
Other: Coarse emulsion — Emulsion is made up of distilled water, olive oil and emulsifier. Emulsion will be flavored, sweetened (sucralose) and served in a portion of 300ml and approximately 3 slices of white bread (50g of available carbohydrate). Additional glass of plain water will be provided with every treatment.
  Arms: Coarse emulsion
Other: Control — Beverage is made up of distilled water and olive oil. Beverage will be flavored, sweetened (sucralose) and served in a portion of 300ml and approximately 3 slices of white bread (50g of available carbohydrate). Additional glass of plain water will be provided with every treatment.
  Arms: Control

SUMMARY:
The aim of this study is to compare the effects of emulsification and lipid droplet size on gastric emptying rate, and to determine if the change in gastric emptying rate can in turn influence postprandial glycemic, insulinemic and lipidemic responses.

DETAILED DESCRIPTION:
This study will be conducted using a randomized, crossover design with three dietary phases: 1) fine emulsion beverage (small lipid droplet size), 2) coarse emulsion beverage (large lipid droplet size) and 3) non-emulsified oil and water. All treatments will be consumed together with bread. All participants will be randomly allocated to the three test meals. Fifteen to twenty participants aged between 21 and 50 years will be recruited from the general public in Singapore.

During the testing sessions, participants' glycemic, insulinemic, lipidemic responses and gastric emptying to the test meals will be measured. Gastric antral distention ultrasound measurement is an indirect measure of gastric emptying rate. Participants' metabolic satiety for the test meals will also be assessed at regular intervals throughout the testing session. Each testing session will take approximately four hours in duration and the testing sessions will take place at least five days apart.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese male subjects aged between 21 and 50 years
* Body mass index between 20.0 to 24.9 kg/m2
* Normal blood pressure (<140/90 mmHg)
* Fasting blood glucose <6.0 mmol/L

Exclusion Criteria:

* People with major chronic disease such as heart disease, cancer or diabetes mellitus
* People with family history of diabetes or familial cholesterolaemic
* People with history of liver or renal problems
* People who have intolerances or allergies to test products
* Individuals who are taking insulin or drugs known to affect glucose metabolism and body fat distribution
* People with a major medical or surgical event requiring hospitalization within the preceding three months
* Individuals with the presence of disease or drugs which influence digestion and absorption of nutrients

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Glycemic response | 4 hours post-prandial (0, 15, 30, 45, 60, 90, 120, 150, 180, 210 and 240 min)
  Blood glucose response to the test meal measured over 4 hours

SECONDARY OUTCOMES:
Insulinemic response | 4 hours post-prandial (0, 15, 30, 45, 60, 90, 120, 150, 180, 210 and 240 min)
  Plasma insulin response to the test meal measured over 4 hours
Triglycerides response | 4 hours post-prandial (0, 15, 30, 45, 60, 90, 120, 150, 180, 210 and 240 min)
  Plasma triglycerides response to the test meal measured over 4 hours
Non-esterified fatty acid (NEFA) response | 4 hours post-prandial (0, 15, 30, 45, 60, 90, 120, 150, 180, 210 and 240 min)
  Plasma NEFA response to the test meal measured over 4 hours
Gastric emptying | 2 hours post-prandial (0, 15, 45, 90 and 120 min)
  Gastric antrum dimension measured over 2 hours
Post-test-meal subjective appetite rating | 4 hours (0, 15, 30, 45, 60, 90, 120, 150, 180, 210 and 240 min)
  Appetite ratings will be collected after test meal consumption using a previously validated visual analog scales

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore, Singapore